CLINICAL TRIAL: NCT00626808
Title: A Post Marketing Evaluation of the Effectiveness of the Risk Minimization Plan For Use of FluMist Among Children Less Than 5 Years of Age
Brief Title: A Post Marketing Evaluation of the Effectiveness of FluMist Risk Minimization Plan in Children
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Collaborators: RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: MI-MA175
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-07

CONDITIONS: Asthma; Wheezing; Immunosuppression
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Children less than 24 months of age
  Interventions: Drug: No Intervention
- 2: Children 24 to 59 months of age with a claim associated with a diagnosis of asthma
  Interventions: Drug: No Intervention
- 3: Children 24 to 59 months of age without a claim associated with a diagnosis of asthma, but with dispensed medication for wheezing
  Interventions: Drug: No Intervention
- 4: Children 24-59 months of age with immunosuppression
  Interventions: Drug: No Intervention

INTERVENTIONS:
Drug: No Intervention — There were no interventions. No subjects were enrolled in this retrospective database study.

SUMMARY:
This is a retrospective cohort study of children included in a large medical insurance claims database.

DETAILED DESCRIPTION:
* To evaluate the rate of FluMist administration compared to other influenza vaccine use in the following pediatric populations:

  * Children younger than 24 months of age
  * Children 24-59 months of age with a claim associated with a diagnosis of asthma
  * Children 24-59 months of age without a claim associated with a diagnosis of asthma, but with dispensed medication for wheezing
  * Children 24-59 months of age with immunosuppression
* To describe, in children in the above populations who receive FluMist, the type and number of Emergency Room visits or hospitalizations associated with an insurance claim within 42 days of receiving FluMist
* To explore the rationale for FluMist immunization of pediatric populations that are excluded from recommended usage by characterizing the use in these populations

ELIGIBILITY:
* Children less than 24 months of age during August through January/February.
* Children <24 to 59 months of age during August through January/February, with:

  * two outpatient claims for asthma, or
  * one inpatient/emergency room claim for asthma, or
  * one outpatient claim for asthma and at least one SABA prescription during a defined 12-month period.
* Children <24 to 59 months of age during August through January/February, without any claims associated with a diagnosis of asthma, but with at least one dispensing for SABA, as indicated by pharmacy claims during a defined 12-month period.
* Children 24 to 59 months of age during August to January/February with evidence of immunosuppression prior to the date of influenza vaccination based on available medical and pharmacy claims.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children < 60 months of age.
Sampling Method: Non-Probability Sample
Enrollment: 321697 (Actual)
Dates: Start 2007-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Ambrose, M.D., Study Director — MedImmune LLC
Locations (1):
- Research Site, Research Triangle Park, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a retrospective descriptive cohort study of participants up to 59 months of age included in a large medical insurance claims database. Participants up to 59 months of age were screened for vaccination with FluMist or TIV as part of routine clinical practice.
Groups:
- Participants Less Than 24 Months of Age: Participants less than 24 months of age
- Participants 24-59 Months of Age With Asthma: Participants 24-59 months of age with a claim associated with a diagnosis of asthma
- Participants 24-59 Months of Age With Wheezing: Participants 24-59 months of age without a claim associated with a diagnosis of asthma, but with dispensed medication for wheezing
- Participants 24-59 Months of Age With Immunosuppression: Participants 24-59 months of age who had claims associated with any of the following: transplantation, congenital immune deficiency, symptomatic human immunodeficiency virus, hematologic/lymphatic malignancy; immunosuppressive therapy other than systemic corticosteroids within the previous 16 weeks; systemic corticosteroids
Period: Overall Study
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Started | 254464 | 34316 | 30011 | 2906
Completed | 254464 | 34316 | 30011 | 2906
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression | Total
Number analyzed (Participants) | 254464 | 34316 | 30011 | 2906 | 321697
Age, Customized [Number; unit: children]
  < 24 months | 254464 | 0 | 0 | 0 | 254464
  >= 24 months | 0 | 34316 | 30011 | 2906 | 67233
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was not collected for this database study.
  Participants
    Female | NA — Gender was not collected from database. | NA — Gender was not collected from database. | NA — Gender was not collected from database. | NA — Gender was not collected from database. | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — Gender was not collected from database. | NA — Gender was not collected from database. | NA — Gender was not collected from database. | NA — Gender was not collected from database. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: FluMist Use in Participants up to 59 Months of Age
Description: Among participants up to 59 months of age who received any flu vaccine, number who received FluMist
Time Frame: 2009-2010
Population: General population of participants aged < 24 months, participants 24-59 months with asthma, participants 24-59 months with wheeing, and participants 24-59 months with immunosuppression.
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 254464 | 34316 | 30011 | 2906
Number of participants | 775 | 3457 | 5821 | 361

2. Primary Outcome: Vaccinating Physician Specialty: Pediatrician or Pediatric Specialist
Description: Specialty of vaccinating physician who provided FluMist.
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of physicians
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of physicians | 553 | 2782 | 4704 | 291

3. Primary Outcome: Vaccinating Physician Specialty: General/Family Practitioner
Description: Specialty of vaccinating physician who provided FluMist
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of physicians
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of physicians | 60 | 140 | 267 | 13

4. Primary Outcome: Vaccinating Physician Specialty: Other
Description: Specialty of vaccinating physician who provided FluMist
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of physicians
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of physicians | 103 | 346 | 581 | 37

5. Primary Outcome: Vaccinating Physician Specialty: Unknown
Description: Specialty of vaccinating physician who provided FluMist
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of physicians
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of physicians | 59 | 189 | 269 | 20

6. Primary Outcome: Geographic Region: Northeastern
Description: Geographic region of parents' residence among participants receiving FluMist
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 64 | 353 | 392 | 20

7. Primary Outcome: Geographic Region: North Central
Description: Geographic region of parents' residence among participants receiving FluMist
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 214 | 755 | 1635 | 101

8. Primary Outcome: Geographic Region: Southern
Description: Geographic region of parents' residence among participants receiving FluMist
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 364 | 1937 | 3127 | 204

9. Primary Outcome: Geographic Region: Western
Description: Geographic region of parents' residence among participants receiving FluMist
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 132 | 404 | 662 | 36

10. Primary Outcome: Number of Outpatient Visits: 0
Description: Among participants vaccinated with FluMist, the number who had 0 outpatient visits in the 3 months prior to vaccination
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 147 | 910 | 1994 | 61

11. Primary Outcome: Number of Outpatient Visits: 1
Description: Among participants vaccinated with FluMist, the number who had 1 outpatient visit in the 3 months prior to vaccination
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 246 | 987 | 1724 | 99

12. Primary Outcome: Number of Outpatient Visits: 2 or More
Description: Among participants vaccinated with FluMist, the number who had 2 or more outpatient visits in the 3 months prior to vaccination
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 382 | 1560 | 2103 | 201

13. Primary Outcome: Number of Days With a Respiratory Claim in 28 Days Prior to Vaccination: 0
Description: Among participants vaccinated with FluMist, the number of days with a respiratory claim (asthma, acute respiratory distress, bronchospasm, influenza, respiratory syncytial virus, bronchiolitis, bronchitis, pneumonia, croup, sinusitis, adenovirus infection, coxsackie virus infection, rhinovirus infection, nasopharyngitis, laryngitis and tracheitis, upper respiratory infection, cough) in the 28 days prior to vaccination.
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 677 | 2778 | 5049 | 245

14. Primary Outcome: Number of Days With a Respiratory Claim in 28 Days Prior to Vaccination: 1
Description: as for outcome 13
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 95 | 670 | 769 | 114

15. Primary Outcome: Number of Days With a Respiratory Claim in 28 Days Prior to Vaccination: 2 or More
Description: as for outcome 13
Time Frame: 2009-2010
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Participants Less Than 24 Months of Age | Participants 24-59 Months of Age With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Number analyzed (Participants) | 775 | 3457 | 5821 | 361
Number of participants | 3 | 9 | 3 | 2

ADVERSE EVENTS:
Time Frame: 2009-2010
Description: This retrospective database study examined claims for hospitalizations or emergency department visits within 42 days after claims for influenza vaccination. No participants were entered in the study and no investigational product was administered.
Arm/Group | Participants Less Than 24 Months of Age | Children 24-59 Months With Asthma | Participants 24-59 Months of Age With Wheezing | Participants 24-59 Months of Age With Immunosuppression
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it is understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.